CLINICAL TRIAL: NCT07068022
Title: Development and Validation of an Obstetric Organ Dysfunction Score to Predict Mortality in Intensive Care Unit: A Multicenter, Prospective, Cohort Study
Brief Title: Organ Dysfunction Score for Obstetric Patients
Acronym: SOFA-OBS
Status: Not yet recruiting | Type: Observational
Sponsor: Daniela Vasquez (Other)
Responsible Party: Sponsor-Investigator, Daniela Vasquez, Medical Doctor, Researcher, Argentinian Intensive Care Society
Organization: Argentinian Intensive Care Society (Other)
Other Study IDs: PRIISABA 15646
Record Dates: First submitted 2025-06-28; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy; Postpartum; Organ Dysfunction; Critical Care, Intensive Care; Sepsis
Keywords: Sequential Organ Failure Assessment score; Pregnancy; Postpartum; Critical care; Intensive Care Unit; Creatinine; Peripheral oxygen saturation; Hypotension; Maternal mortality; Mortality; Sepsis; Septic shock; Multicenter study
MeSH Terms: conditions — Sepsis; Hypotension; Maternal Death; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obstetric patients= pregnant and postpartum (< 3 days) patients requiring ICU admission: All pregnant and postpartum (< 3 days) patients requiring ICU admission will be followed during their ICU-LOS. The predictive validity for ICU mortality of an adjusted to obstetric patients Sequential Organ Failure Assessment (SOFA-OBS) score will be compared to the predictive validity of a non-modified Sequential Organ Failure Assessment (SOFA) score.
  Interventions: Other: Organ dysfunction score adjusted to obstetric patients (SOFA-OBS)

INTERVENTIONS:
Other: Organ dysfunction score adjusted to obstetric patients (SOFA-OBS) — The obstetric SOFA (SOFA-OBS) adjusts renal and cardiovascular variables to physiological changes of pregnancy. Moreover, it simplifies respiratory evaluation, in terms of replacing arterial blood gases (ABG) for peripheral oxygen saturation/fraction of inspired oxygen (spO2/FiO2), when ABGs were not available. Variables unchanged during pregnancy (neurologic, hepatic and platelets), won't be modified.

SUMMARY:
The goal of this observational study is to develop and evaluate an organ dysfunction score adapted to pregnancy and early puerperium (SOFA-OBS) that also incorporates a non-invasive tool to evaluate respiratory function (pulse oximeter).

The main question it aims to answer is: Does an organ dysfunction score adapted to pregnant and postpartum patients have a higher capacity to predict mortality than a non-adjusted organ dysfunction score? Participants: Patients requiring ICU (Intensive Care Units) admission, who are either pregnant or postpartum (up to 3 days after giving birth). The investigators aimed to include 130 participants.

The investigators will only collect participants' data and laboratory results that ICU doctor usually need for clinical practice. No additional interventions are required. Moreover, the investigators will evaluate if measuring participants' oxygenation through a non-invasive tool (pulse oximeter) is equally effective as measuring oxygenation by an arterial puncture.

Background: When managing severely ill patients in ICU, the investigators often use what it is called scores. Scores refer to a numerical value assigned to a patient's condition, which often predict outcome. The Sequential Organ Failure Assessment (SOFA) score is a scoring system that assess severity of organ dysfunction (in liver, kidney, blood pressure, respiratory, neurologic and platelets). It also identifies patients with severe infections (sepsis) and patients with bad outcomes.

Patients undergoing pregnancy or early postpartum develop physiological changes, such us a decrease in creatinine (a laboratory test measuring kidney function) and a decrease in blood pressure during the second trimester. These changes are not considered by the SOFA score. Actually, there is not an organ dysfunction score adapted to pregnant/postpartum patients to be used in the ICU. Moreover, a blood sample taken by arterial puncture is required to evaluate respiratory function by the SOFA score, which is a painful procedure. Instead, the investigators could evaluate respiratory function using a pulse oximeter, which measures peripheral oxygen saturation without needing an arterial puncture.

Potential benefits: A SOFA-OBS would hopefully become a more precise tool than general SOFA to evaluate organ dysfunction and to predict outcome among these patients. It would also help to detect sepsis earlier and treat it promptly, which might help reducing its mortality.

DETAILED DESCRIPTION:
INTRODUCTION The Sequential Organ Failure Assessment (SOFA) score was initially developed in a consensus meeting organized by the European Society of Intensive Care in 1996. The aim of the score was to quantify and objectively describe the degree of organ dysfunction or failure in critically ill patients (1). The SOFA score describes a continuum process from normality to dysfunction and failure for six organ systems (respiratory, hematologic, hepatic, cardiovascular, neurologic and renal) (1). Although primary objective of SOFA score was descriptive, numerous studies have proven its prognostic value as well. There is a strong association between SOFA, number of dysfunctions upon admission and SOFA trends in the first 48h and ICU mortality (2, 3).

The SOFA score is a key component of the last definition of sepsis. In 2016, the European Society of Critical Care and the American Society of Critical Care developed and validated a new definition of sepsis. Sepsis was then considered as a life-threatening organ dysfunction caused by a dysregulated host response to infection (3). SOFA score was chosen to identify organ dysfunction due to its simplicity and widespread use. Organ dysfunction was defined as a change in total SOFA score of ≥ 2 points (3). This definition was validated by many studies of different countries, including Argentina (4, 5).

The SOFA score was developed and validated in a population of adult critically ill patients. Thus, its calibration for other populations with particular physiological changes, such as children or obstetric patients, could be inadequate. While some scores, like the PELOD (6, 7) or modified SOFA (8) were developed and validated for pediatric patients, there is no one suitable for obstetric patients yet. General SOFA score was associated with mortality among obstetric patients (9-12) but its predictive validity could be improved if adjustments to pregnancy were performed. Although two groups proposed modified SOFA scores adjusted to obstetric patients, these scores presented clear deficiencies and were not validated (13, 14). The development of an adjusted and calibrated organ dysfunction score for obstetric patients, would improve the validity of the score to predict ICU mortality, and would provide a reliable tool to be incorporated into the definition of maternal sepsis (15, 16). Obstetric sepsis account for 11% of global maternal mortality and for 19%, when abortion-related deaths are added, as most of them are due to sepsis (17). Developing a validated instrument to define sepsis in this population, would improve its recognition and would eventually promote its early treatment, which is associated with better outcomes (18).

Barriers for using the non-adjusted SOFA score to diagnose sepsis in obstetric patients are mainly related to renal and cardiovascular systems. SOFA score sets a creatinine of ≥1.2 mg/dl as the lower cut-off point to identify kidney dysfunction (1). However, pregnant patients and those in early puerperium, present an increased in cardiac output, in renal plasma flow and in glomerular filtration rate, which in turn decrease normal creatinine levels to <0.9 mg/dl in any trimester of pregnancy (19, 20) and in the first 2 weeks postpartum (20-22). Thus, a non-adjusted SOFA score underestimates renal dysfunction in obstetric patients. In terms of cardiovascular dysfunction, mean arterial pressure (MAP) normally decreases during the second trimester of pregnancy, up to approximately 65 mmHg. However, for the general SOFA score any value of MAP ≤70 mmHg is considered abnormal, which will overestimate hemodynamic dysfunction during that trimester (1). In addition to the abovementioned required adjustments, respiratory evaluation of SOFA is usually lacking among obstetric patients. This evaluation is performed through the paO2/FiO2 ratio, which requires an arterial blood gas (ABG) extraction (23, 24). ABG measurement could be unavailable in some low-resource settings, but also could be missing due to a deliberate physician decision of avoiding arterial gas extraction in these patients (24). Using the relationship between the peripheral oxygen saturation over the inspired fraction of oxygen (spO2/FiO2) could address this deficiency. The spO2/FiO2 ratio is a validated, widely available and non-invasive surrogate of paO2/FiO2 ratio to evaluate respiratory performance (25, 26). The use of a paO2/FiO2 ratio surrogate, such as the spO2/FiO2, improves SOFA score specificity compared to the decision of considering the missing value as normal (24) and it is a key factor when SOFA score is used to define sepsis (15).

The main objective of this study is to develop and validate an organ dysfunction score adjusted to obstetric patients (SOFA-OBS) to predict ICU mortality among pregnant and early postpartum patients requiring ICU admission.

I. Background and significance There were two previous attempts to adapt the SOFA score to the obstetric population. In 2016, Blanco Esquivel et al. (13), developed a SOFA score adjusted to obstetric patients; however, the variable chosen to be modified was questionable. The authors proposed lowering normal cut-off point for paO2/FiO2 and SaO2/FiO2, assuming pregnant patients have lower paO2 levels due to a decreased total lung capacity (TLC). However, pregnant patients neither present a reduction in TLC nor a decrease in oxygenation; thus, SOFA score cut-off values for respiratory evaluation should not be modified (27). Moreover, pregnancy renal and hemodynamic changes were not considered. In 2017, the Society of Obstetric Medicine of Australia and New Zealand proposed an obstetric SOFA. This score removed scores of 3 and 4 in each category for simplification and reduced creatinine cut-off point to 1 mg/dl (14). However, this creatinine value is still higher than the expected for obstetric patients. In addition, no adjustments were done for MAP during the second trimester and no validation of the modified obstetric SOFA was performed.

The SOFA-OBS score proposed in this study would be the first adjusting creatinine and MAP to the obstetric population in a prospective and multicenter study, using the best evidence available (28, 29). In addition, it would be the first study evaluating SpO2/FiO2 calibration among these patients, which might improve the specificity and predictive validity of the score. The development and validation of an obstetric SOFA score to be used in the diagnose of maternal sepsis, would contribute to its early recognition and prompt treatment, which instead would hopefully reduce maternal mortality associated with sepsis.

II. Objectives

Primary objective:

- To develop an obstetric SOFA score (SOFA-OBS) adjusted to physiological changes of pregnancy and to validate the SOFA-OBS during the first 24h in ICU (SOFA-OBS24h) to predict ICU mortality among obstetric patients.

Secondary Objectives:

* To validate the SOFA-OBS to predict maternal sepsis among obstetric patients requiring ICU admission
* To validate SOFA-OBS to predict sepsis associated mortality among obstetric patients requiring ICU admission
* To evaluate the mean SOFA-OBS (SOFA-OBS mean) to predict mortality among obstetric patients requiring ICU admission
* To evaluate the maximum SOFA-OBS (SOFA-OBS max) to predict mortality among obstetric patients requiring ICU admission
* To evaluate the impact of SOFA-OBS trend during the first 48 h in ICU (SOFAΔ48) (increase, decrease, no changes) on ICU mortality
* To evaluate the relationship between the presence of each organ dysfunction/failure during the first 24h in ICU and ICU mortality
* To evaluate the relationship between the number of organ dysfunctions/failures during the first 24h in ICU and ICU mortality
* To evaluate the validity of the conventional septic shock definition (15) to predict mortality among obstetric patients admitted to ICU using the SOFA-OBS to define dysfunction
* To evaluate the validity of the second trimester septic shock definition (2T-SS) to predict ICU mortality among obstetric patients using the SOFA-OBS to define dysfunction

Null Hypothesis:

* SOFA-OBS does not have higher predictive validity for ICU mortality among obstetric patients requiring ICU admission than non-adjusted SOFA

Alternative Hypothesis:

- SOFA-OBS has higher predictive validity for ICU mortality among obstetric patients requiring ICU admission than non-adjusted SOFA

III. Material y Methods This study will consist in a development phase and a validation phase of an obstetric SOFA (SOFA-OBS). The investigators will follow TRIPOD (Transparent Reporting of a multivariable prediction model for Individual Prognosis or Diagnosis) guidelines and TRIPOD check-list (30). Following, investigators describes elements not covered elsewhere.

Sample size calculation:

The sample size was estimated considering the main objective, which includes validity assessment of an organ dysfunction score modified to obstetric patients (SOFA-OBS), through the AUROC. The investigators considered information published by Oliveira Neto et al. (31), which reports an obstetric mortality of 2.6% in a 673 patients cohort. In order to detect an AUROC of 0.9, an alpha error of 5% and a power of 80%, 130 patients are required (4 presenting the outcome and 126 not presenting it). Statistical package pROC of the statistical software R was used to calculate sample size.

Theoretical and operational variables definitions:

Outcome variables:

1. Obstetric patients ICU mortality: defined elsewhere. This outcome cannot be blinded to in site researchers; however, it is a definite outcome, not requiring any interpretation. Moreover, the final data analysis will be performed by a separate team from the one collecting them.
2. Sepsis-related obstetric ICU mortality: defined elsewhere Although ICU mortality is an objective outcome, as previously mentioned, the attribution of sepsis as cause of death requires some interpretation. This outcome variable cannot be blinded, but the investigators will use an accepted and concise definition supported by objective variables, such as a change in SOFA score of at least 2 points and a suspected infection triggering cultures or antibiotics administration. The final data analysis will be performed also by a separate team from the one collecting data.

Predictor variables:

1. Sequential Organ Failure Assessment (SOFA) and modified SOFA scores (obstetric SOFA: SOFA-OBS):

   The investigators decided to adapt the Sequential Organ Failure Assessment (SOFA) score to the obstetric population. The SOFA score is used worldwide and is simple. It also has high predictive validity for mortality among critically ill patients in general and critically ill obstetric patients, in particular. However, it was not calibrated for obstetric patients.

   The SOFA score is a key component of last sepsis definition (15). Although sepsis is an important cause of maternal mortality, a SOFA score adjusted to obstetric patients, which could be incorporated in sepsis definition, is still unavailable.

   SOFA score will be measured according to its original version. Six organ systems (respiratory, hematologic, hepatic, cardiovascular, neurologic and renal) are evaluated (1). The worst value for each organ on a day is recorded and a score of 0 to 4 is assigned to each value according to predefined ranges (1, 2). Normal values are assigned 0 points and abnormal values are assigned 1 to 4 points (from least to most abnormal); where 1 and 2 represents organ dysfunction and 3 and 4 represents organ failure (2). Total SOFA score is the results from the sum of the score of each organ (1, 2).

   The obstetric SOFA (SOFA-OBS) adjusts renal and cardiovascular variables to physiological changes of pregnancy. Moreover, it simplifies respiratory evaluation, in terms of replacing arterial blood gases (ABG) for peripheral oxygen saturation/fraction of inspired oxygen (spO2/FiO2), when ABGs were not available. Variables unchanged during pregnancy (neurologic, hepatic and platelets), won't be modified.

   Organ evaluation according to SOFA and SOFA-OBS score:
   * Neurologic: will be performed through the Glasgow Coma Scale (GCS) (32). If the patient is under sedation, the GCS before sedation (assumed) will be used (3). Should this data be unavailable, GCS recorded will be recorded at 15 (normal) (ECG= 15).
   * Hepatic: will be assessed by measuring total bilirubin levels, as for the original SOFA, because they do not change with pregnancy (19).
   * Hematologic: will be evaluated according to platelet counts, using the same ranges as those from the original SOFA, because platelets count during most pregnancy period are normally ≥150000/mm3, which is the lower cut-off point for the SOFA score (19).
   * Renal: will be assessed with creatinine adjusted to normal changes of pregnancy and early puerperium. Creatinine will be considered abnormal at a cut-off point of ≥0.9 mg/dl (79.58 umol/l), according to data from a systematic review (28), population studies of different regions (20, 21, 33-35) and consensus from general practice (19). The investigators consider this value unifies values described in the literature, decreases false positives and increments specificity.
   * Cardiovascular: for the first and third trimesters of pregnancy, normal mean arterial pressure (MAP) is the same as that of the general population. So, original SOFA cut-off point of abnormality (MAP <70 mmHg) will be considered. During the second trimester, MAP usually descends, thus, cut-off point of abnormality and consequently a SOFA score= 1, will be taken at a MAP of < 65 mmHg, according to Meah and col. metanalysis (29).
   * Respiratory: for patients with arterial blood gases available (ABG) the worst value of arterial partial pressure of oxygen/ fraction of inspired oxygen (paO2/FiO2) ratio will be taken. When ABGs were unavailable, the worst value of pulse oximetry saturation/fraction of inspired oxygen (spO2/FiO2) ratio will be considered, following previously proposed ranges (24, 36).
   * For spO2/FiO2 measurements normal oximetry readings should be ensured. This requires: no position changes neither aspiration 10 minutes before measurement and no changes in ventilatory setting 30 minutes before measurement (26).

   SOFA will be recorded daily, taking the worst value of each parameter (from 0 to 4). Daily total SOFA will represent the sum of the 6 parameters (0-24)(2). Measurements will be taken daily, as far as the patient is pregnant or ≤3 days postpartum, during the whole ICU-LOS and up to discharge or dead.

   The investigators will specifically measure:

   • SOFA24h: SOFA during the first 24h in the ICU
   * SOFAmax: maximum SOFA during ICU-LOS
   * SOFAprom: mean SOFA during ICU-LOS
   * SOFAΔ48: difference between SOFA at 48 h from admission and SOFA on admission
2. Sepsis: the following parameters will be recorded on admission and at any point during ICU-LOS .2.1 Sepsis: life-threatening organ dysfunction caused by a dysregulated host response to infection (15).

2.2 Organ dysfunction: acute change in total SOFA score of ≥ 2 puntos as a result of an infection. A previous SOFA is assumed to be 0 in a patient with no preexistent infection (15).

2.3 Suspected infection: condition requiring cultures order and/or antibiotic onset (15).

2.4 Septic shock: sepsis with persistent hypotension requiring vasopressors to maintain MAP > 65 mmHg and having a serum lactate level > 18 mg/dl (> 2 mmol/L) despite adequate volume resuscitation (15). This definition applies without modifications in pregnant patients during their first or third trimesters, because no changes in MAP are observed at these two points, compared to non-pregnant population.

2.5 Septic shock in the second trimester (SS-2T): sepsis with persistent hypotension requiring vasopressors to maintain MAP > 60 mmHg and having a serum lactate level > 18 mg/dl (> 2 mmol/L), despite adequate volume resuscitation.

Septic shock definition for the general ICU population considers hypotension when MAP persists < 65 mmHg requiring vasopressors, while SOFA score considers hypotension when MAP <70 mmHg. In order to preserve consistency, for septic shock definition during the second trimester, hypotension will be considered when MAP <60 mmHg, while SOFA-OBS score will define hypotension (SOFA= 1) when MAP <60 mmHg.

To blind assessment of predictors for the outcome will be impossible. Investigators collecting SOFA and SOFA-OBS scores will be aware of patients' outcomes (mortality). In order to avoid classification bias, predictive variables will be defined in the same way by all centers, using objective and clear criteria. Moreover, investigators will be asked to record raw data for SOFA components, instead of the scoring itself. The REDcap system will calculate the score for each parameter and the total SOFA score, according to predefined criteria.

Rest of variables that will be collected for the study at each center:

1. Hospital general data:

   a. Localization b. Third level center c. Type of health care: public-private- social security d. Total bed number e. 24h obstetrician available f. Total number of births per year g. High-risk pregnancy care h. Neonatology unit i. 24h anesthesiologist available j. Type of ICU: general, obstetric k. 24 h board certified or trained in critical care physician: l. ICU bed number m. General ICU admissions per year (Mean ± SD) and total number of ICU admissions during the study period n. Obstetric ICU admissions per year (Mean ± SD) and total number of obstetric ICU admissions during the study period
2. Patients' data:

   1. Age
   2. Source of admission to ICU: emergency department, ward, operating room, other hospital)

   <!-- -->

   1. Comorbidity, measured with the Charlson Comorbidity Index (CCI) (37). Causes of admission to ICU: obstetric (occurring only in pregnant/postpartum patients) vs. non obstetric (also occurring in nonpregnant patients) (10).
   2. Specific diagnoses of admission
   3. Obstetric history:

   i. Gestational age on admission to ICU (weeks) ii. Gestational age on admission classified in trimesters (29): i. First trimester: 6-13 weeks ii. Second trimester: 14-27 weeks iii. Third trimester: ≥28 weeks iii. Parity. iv. Prenatal care v. Should pregnancy terminate during ICU-LOS: gestational age at termination will be recorded as well as fetal/neonatal outcome.

   d. ICU data: i. Severity of illness during the first 24 h in ICU through the Simplified Acute Physiologic Score (SAPS II) (38) ii. ICU interventions: advanced respiratory support (high Flow nasal cannula [HFNC], Non-invasive ventilation [NIV], invasive mechanical ventilation [IMV]); renal replacement therapy (RRT) and hemodynamic monitoring.

   iii. Documented infection in ICU: Yes, No; type of infection (pneumonia, urinary tract infection, catheter related bacteremia, bacteriemia of unknown source, endometritis, septic abortion, chorioamnionitis, surgical site infection.

   e. Additional outcome variables: i. Total number of livebirths during the study period. ii. ICU-length of stay (ICU-LOS). iii. Hospital-LOS. iv. Additional mortality data: i. Maternal mortality rate (MMR): is defined as female deaths from any cause related to or aggravated by pregnancy or its management, occurring during pregnancy or within 6 weeks of termination of pregnancy, irrespective of the duration and site of the pregnancy, for a specific period of time and expressed over 100000 live births (17). The investigators will adapt this definition, as only pregnant patients or those in their early puerperium (up to 3 days after birth) will be included in this study Maternal mortality ratio will be defined for this study as: Non-surviving obstetric patients admitted to ICU during the study period/ number of live births among the same population during the same study period.

   ii. MMR associated with direct causes= non-surviving obstetric patients admitted to ICU for a direct cause during the study period/ number of live births among the same population during the same study period.

   iii. MMR associated with indirect causes= non-surviving obstetric patients admitted to ICU for an indirect cause during the study period/ number of live births among the same population during the same study period.

   ii. Hospital mortality: i. Obstetric patient hospital mortality: Number of obstetric patients who required ICU admission during the study period and did not survive at hospital discharge/ all obstetric patients who required ICU admission during the study period.

   iii. Pregnancy outcomes i. Termination of pregnancy during ICU-LOS: Yes/No 1. Gestational age at termination of pregnancy (39)=
   1. Term: ≥ 37 weeks
   2. Preterm: < 37 weeks

   i. Extrem preterm: 22-27+6 weeks ii. Early preterm: 28-31+6 weeks iii. Late preterm: 32-36 +6 weeks ii. Discharged pregnant iv. Fetal/neonatal outcomes: i. Survivors: both livebirths and discharged pregnancies will be included in this category/total number of obstetric patients admitted to the ICU during the study period.

   ii. Non survivors: both spontaneous abortions and perinatal deaths will be included in this category/ total number of obstetric patients admitted to the ICU during the study period: 1. Spontaneous abortions: those occurring < 22 weeks 2. Perinatal deaths: fetal (≥ 22 weeks) and early neonatal deaths (0-6 days after birth) (39).

   IV. Handling missing data The investigators will set Redcap with required fields, which will not allow researchers to continue filling forms if data is lacking. In addition, a research assistant will check the database weekly in order to look for missing or incongruent data, contacting local researchers to complete or review data. To avoid bias related to potential missing data, while assuming it is missing at random, primary objective analysis will be replicated after multiple imputations.

   V. Statistical analysis Categorical variables will be presented as numbers (%) and continuous variables as mean ± SD or median [IQR], according to their distribution. The Shapiro-Wilk test will determine whether data is normally distributed or not. Categorical variables will be presented as number and percentage (%). Normally distributed continuous variables will be compared with Student t-test and non-normally distributed continuous data with Wilcoxon test. Categorical variables will be compared with chi-square or Fisher test. Multiple comparisons of parametric, non-parametric and categorical variables will be analyzed with one factor ANOVA, Kruskal Wallis o multiple chi-square tests, respectively.

   SOFA-OBS predictive validity for ICU mortality will be evaluated through its capacity to distinguish survivors from non-survivors (discrimination) and through the agreement between observed and predictive probabilities of death (calibration). Discrimination will be assessed by the area under the receiver operating characteristic curve and its 95% confidence interval (AUROC IC 95%) and calibration by the Hosmer-Lemeshow statistics. The same analysis will be repeated for the general SOFA score. Finally, both scores (SOFA-OBS and SOFA) performances will be compared by AUROC and c-index. Predictive validity for mortality of each organ dysfunction, measured by maximum SOFA of each organ, will be assessed by AUROC. Bootstrapping will be used for internal validation.

   The relation between the presence of organ dysfunction/failure during the first 24h in ICU and ICU mortality will be assessed through Chi2 test, measuring the percentage of non-survivors among all patients presenting each category of organ dysfunction/failure. Creatinine cut-off points for each SOFA score category to predict ICU mortality will be determine using Fisher algorithm to obtain ordinal variables with k +1 categories. The relation between trends in SOFA score during the first 48h (increase, decrease, no change) and ICU mortality, will be assessed through Chi2 multiple test.

   Predictive validity of mortality of a change in SOFA-OBS ≥2 among obstetric patients with suspected infection in the ICU will be assessed through AUROC and its 95% CI. This analysis will be repeated for general SOFA score and both results will be compared.

   The relationship between predictive and outcome variables, will be evaluated through multivariate analysis, adjusting for potential confounders. A p value <0.05 will be considered significant. SPSS20 will be used for data analysis.

   VI. Procedures and tools for collecting data and data quality control

   Data for this study will be collected as part of standard care in the ICU. In the case the patient does not require daily laboratory, data will be record as missing.
   1. Tools for collecting data: the same case report form (CRF) will be used across all centers. Data will be collected through REDCap.
   2. Data quality control: variables will be clearly defined in the manual of procedures, to ensure data validity. Data will be initially validated and audited by REDCap in terms of mistakes associated with typing or normal ranges. A research assistant will perform a weekly database monitoring, looking for data consistency and quality. If any inconsistency, error or missingness are detected, local researchers will be contacted to correct or fill them. Predetermined virtual meetings will be arranged for training and addressing queries. All sites will use the same definitions for variables. Local investigators will be asked to insert raw data into REDCap and the system will calculate different scores (e.g. SAPS II, SOFA, etc.).

   VII. Ethical considerations in human research and informed consent This is an observational study using data normally collected for clinical practice. The study was approved by the institutional review board of the Argentinian Society of Critical Care Medicine (Identifier PRIISABA-15646). As the study is also prospective, informed consent will be obtained before enrolling participants. The study will be performed in accordance with ethical standards laid down in the 1964 Declaration of Helsinki and later amendments and with national and regional guidelines for research in human beings (Argentinian National Ministry of Health-Res. 1480/2011 and Law for protecting rights of participants in Health Research 3301/2009 of the city of Buenos Aires, respectively). Each participant site, will obtain approval from their IRB and will follow their requirements. The organizer site will get a copy of the IRB approval from each center.

   Confidentiality and privacy will be protected according to the Argentinian National Law 25326 for Protecting personal data. Each site and patient will get a code number to keep anonymity. No personal data will be inserted into REDcap.

ELIGIBILITY:
Inclusion Criteria:

All of the following=

* Pregnant (at any gestational age) or post-partum patients (at ≤3 days postpartum)
* ≥ 18 years old
* Requiring admission to ICU for any reason
* Staying in the ICU for ≥ 24h
* Giving her consent to participate. Patients will be recruited consecutively until reaching the sample size.

Exclusion Criteria:

Any of the following=

* Patients <18 years old
* Non-pregnant patients
* ≥ 4 days postpartum
* Patients or surrogates not giving consent to participate
* ICU-LOS < 24 h

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in ICUs from third level hospitals from Latin American countries.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Obstetric patients ICU mortality | From patient enrollment to patient discharge from ICU (alive/dead) or 28-days post-enrollment, whichever occur first.
  Non-surviving obstetric patients admitted to ICU during the study period/ all obstetric patients admitted to ICU during the same period
Sepsis-related obstetric ICU mortality | From patient enrollment to patient discharge from ICU (alive/dead) or 28-days post-enrollment, whichever occur first.
  Non-surviving obstetric patients admitted to ICU during the study period, presenting sepsis on admission or developing sepsis during their ICU-LOS/All obstetric patients admitted to ICU during the same period, presenting sepsis on admission or developing sepsis during their ICU-LOS

CONTACTS AND LOCATIONS:
Overall Officials: Daniela N. Vasquez, MD, Principal Investigator — Sanatorio Anchorena Recoleta
Locations (17):
- Argentina (14):
  - Sanatorio Itoiz, Avellaneda, Buenos Aires
  - Sanatorio Anchorena Recoleta, City of Buenos Aires, Buenos Aires
  - Hospital Simplemente Evita, González Catán, Buenos Aires
  - Hospital Mi Pueblo Florencio Varela, San Juan Bautista, Buenos Aires
  - Hospital Thompson, San Martín, Buenos Aires
  - Sanatorio Anchorena San Martín, San Martín, Buenos Aires
  - Hospital Materno Infantil Dr. F Escardó, Tigre, Buenos Aires
  - Hospital de la Madre y el Niño, La Rioja, La Rioja Province
  - Hospital Regional Diego Paroissien, Mendoza, Mendoza Province
  - Maternidad Provincial Teresita Baigorria, San Luis, San Luis Province
  - Hospital Regional Ramón Carrillo, Santiago del Estero, Santiago del Estero Province
  - Sanatorio Antártida, City of Buenos Aires
  - Sanatorio Finochietto, City of Buenos Aires
  - Sanatorio Guemes, City of Buenos Aires
- Hospital Gineco Obstétrico Isidro Ayora, Quito, Ecuador
- Hospital Materno Infantil 1 de mayo, San Salvador, El Salvador
- Hospital de Clínicas Dr. Manuel Quintela, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No
We would have like to share IPD, now we know its significance. Unfortunately, at the moment we invited all centers to participate and when the manuscript was sent to the IRB of the Argentinian society of critical care we were not aware of the possibility of sharing IPD. Thus, we did not ask permission from centers neither from the IRB to do so.

REFERENCES:
- [Background] Wolff RF, Moons KGM, Riley RD, Whiting PF, Westwood M, Collins GS, Reitsma JB, Kleijnen J, Mallett S; PROBAST Groupdagger. PROBAST: A Tool to Assess the Risk of Bias and Applicability of Prediction Model Studies. Ann Intern Med. 2019 Jan 1;170(1):51-58. doi: 10.7326/M18-1376. PMID 30596875
- [Background] Oliveira-Neto A, Parpinelli MA, Cecatti JG, Souza JP, Sousa MH. Sequential organ failure assessment score for evaluating organ failure and outcome of severe maternal morbidity in obstetric intensive care. ScientificWorldJournal. 2012;2012:172145. doi: 10.1100/2012/172145. Epub 2012 Feb 14. PMID 22454600
- [Background] Blencowe H, Hug L, Moller AB, You D, Moran AC. Definitions, terminology and standards for reporting of births and deaths in the perinatal period: International Classification of Diseases (ICD-11). Int J Gynaecol Obstet. 2025 Jan;168(1):1-9. doi: 10.1002/ijgo.15794. Epub 2024 Aug 11. PMID 39127912
- [Background] Le Gall JR, Lemeshow S, Saulnier F. A new Simplified Acute Physiology Score (SAPS II) based on a European/North American multicenter study. JAMA. 1993 Dec 22-29;270(24):2957-63. doi: 10.1001/jama.270.24.2957. PMID 8254858
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Schuler A, Wulf DA, Lu Y, Iwashyna TJ, Escobar GJ, Shah NH, Liu VX. The Impact of Acute Organ Dysfunction on Long-Term Survival in Sepsis. Crit Care Med. 2018 Jun;46(6):843-849. doi: 10.1097/CCM.0000000000003023. PMID 29432349
- [Background] Harel Z, McArthur E, Hladunewich M, Dirk JS, Wald R, Garg AX, Ray JG. Serum Creatinine Levels Before, During, and After Pregnancy. JAMA. 2019 Jan 15;321(2):205-207. doi: 10.1001/jama.2018.17948. PMID 30644975
- [Background] Gao Y, Jia J, Liu X, Guo S, Ming L. Trimester-Specific Reference Intervals of Serum Urea, Creatinine, and Uric Acid Among Healthy Pregnant Women in Zhengzhou, China. Lab Med. 2021 May 4;52(3):267-272. doi: 10.1093/labmed/lmaa088. PMID 33145592
- [Background] Agampodi SB, Agampodi TC, Amarasinghe GS, Warnasekara JN, Hettiarachchi AU, Jayasinghe IU, Koralegedara IS, Abeyrathna P, Srimantha S, de Silva FN, Gunarathne SP, Wickramasinghe ND. Serum creatinine and estimated glomerular filtration rate (eGFR) in early pregnancy and changes during the pregnancy. PLOS Glob Public Health. 2023 Jan 26;3(1):e0000443. doi: 10.1371/journal.pgph.0000443. eCollection 2023. PMID 36962935
- [Background] Collins GS, Moons KGM, Dhiman P, Riley RD, Beam AL, Van Calster B, Ghassemi M, Liu X, Reitsma JB, van Smeden M, Boulesteix AL, Camaradou JC, Celi LA, Denaxas S, Denniston AK, Glocker B, Golub RM, Harvey H, Heinze G, Hoffman MM, Kengne AP, Lam E, Lee N, Loder EW, Maier-Hein L, Mateen BA, McCradden MD, Oakden-Rayner L, Ordish J, Parnell R, Rose S, Singh K, Wynants L, Logullo P. TRIPOD+AI statement: updated guidance for reporting clinical prediction models that use regression or machine learning methods. BMJ. 2024 Apr 16;385:e078378. doi: 10.1136/bmj-2023-078378. PMID 38626948
- [Background] Meah VL, Cockcroft JR, Backx K, Shave R, Stohr EJ. Cardiac output and related haemodynamics during pregnancy: a series of meta-analyses. Heart. 2016 Apr;102(7):518-26. doi: 10.1136/heartjnl-2015-308476. Epub 2016 Jan 21. PMID 26794234
- [Background] Wiles K, Bramham K, Seed PT, Nelson-Piercy C, Lightstone L, Chappell LC. Serum Creatinine in Pregnancy: A Systematic Review. Kidney Int Rep. 2018 Oct 29;4(3):408-419. doi: 10.1016/j.ekir.2018.10.015. eCollection 2019 Mar. PMID 30899868
- [Background] Lapinsky SE, Vasquez DN. Acute Respiratory Failure in Pregnancy. Crit Care Clin. 2024 Apr;40(2):353-366. doi: 10.1016/j.ccc.2024.01.005. Epub 2024 Jan 30. PMID 38432700
- [Background] Rice TW, Wheeler AP, Bernard GR, Hayden DL, Schoenfeld DA, Ware LB; National Institutes of Health, National Heart, Lung, and Blood Institute ARDS Network. Comparison of the SpO2/FIO2 ratio and the PaO2/FIO2 ratio in patients with acute lung injury or ARDS. Chest. 2007 Aug;132(2):410-7. doi: 10.1378/chest.07-0617. Epub 2007 Jun 15. PMID 17573487
- [Background] Pandharipande PP, Shintani AK, Hagerman HE, St Jacques PJ, Rice TW, Sanders NW, Ware LB, Bernard GR, Ely EW. Derivation and validation of Spo2/Fio2 ratio to impute for Pao2/Fio2 ratio in the respiratory component of the Sequential Organ Failure Assessment score. Crit Care Med. 2009 Apr;37(4):1317-21. doi: 10.1097/CCM.0b013e31819cefa9. PMID 19242333
- [Background] Schenck EJ, Hoffman KL, Oromendia C, Sanchez E, Finkelsztein EJ, Hong KS, Kabariti J, Torres LK, Harrington JS, Siempos II, Choi AMK, Campion TR Jr. A Comparative Analysis of the Respiratory Subscore of the Sequential Organ Failure Assessment Scoring System. Ann Am Thorac Soc. 2021 Nov;18(11):1849-1860. doi: 10.1513/AnnalsATS.202004-399OC. PMID 33760709
- [Background] Grissom CK, Brown SM, Kuttler KG, Boltax JP, Jones J, Jephson AR, Orme JF Jr. A modified sequential organ failure assessment score for critical care triage. Disaster Med Public Health Prep. 2010 Dec;4(4):277-84. doi: 10.1001/dmp.2010.40. PMID 21149228
- [Background] Hladunewich MA, Lafayette RA, Derby GC, Blouch KL, Bialek JW, Druzin ML, Deen WM, Myers BD. The dynamics of glomerular filtration in the puerperium. Am J Physiol Renal Physiol. 2004 Mar;286(3):F496-503. doi: 10.1152/ajprenal.00194.2003. Epub 2003 Nov 11. PMID 14612381
- [Background] el-Mahallawi MN, el-Din DS, Mahran M, Sabour MS, Fadel HE. Glomerular filtration rate in normal pregnancy and early postpartum period. Obstet Gynecol. 1968 May;31(5):621-6. doi: 10.1097/00006250-196805000-00004. No abstract available. PMID 5646392
- [Background] Legoabe Z, Sebitloane M, Lombard C, Naidoo M, Gray G, Moodley D. Development of normal reference intervals for renal function in pregnancy: a secondary analysis of clinical trial data. J Obstet Gynaecol. 2024 Dec;44(1):2361445. doi: 10.1080/01443615.2024.2361445. Epub 2024 Jun 4. PMID 38832538
- [Background] Abbassi-Ghanavati M, Greer LG, Cunningham FG. Pregnancy and laboratory studies: a reference table for clinicians. Obstet Gynecol. 2009 Dec;114(6):1326-1331. doi: 10.1097/AOG.0b013e3181c2bde8. PMID 19935037
- [Background] Society for Maternal-Fetal Medicine (SMFM). Electronic address: pubs@smfm.org; Plante LA, Pacheco LD, Louis JM. SMFM Consult Series #47: Sepsis during pregnancy and the puerperium. Am J Obstet Gynecol. 2019 Apr;220(4):B2-B10. doi: 10.1016/j.ajog.2019.01.216. Epub 2019 Jan 23. PMID 30684460
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Bonet M, Nogueira Pileggi V, Rijken MJ, Coomarasamy A, Lissauer D, Souza JP, Gulmezoglu AM. Towards a consensus definition of maternal sepsis: results of a systematic review and expert consultation. Reprod Health. 2017 May 30;14(1):67. doi: 10.1186/s12978-017-0321-6. PMID 28558733
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Bowyer L, Robinson HL, Barrett H, Crozier TM, Giles M, Idel I, Lowe S, Lust K, Marnoch CA, Morton MR, Said J, Wong M, Makris A. SOMANZ guidelines for the investigation and management sepsis in pregnancy. Aust N Z J Obstet Gynaecol. 2017 Oct;57(5):540-551. doi: 10.1111/ajo.12646. Epub 2017 Jul 3. PMID 28670748
- [Background] Blanco Esquivel LA, Urbina JM, Zeron HM. Approach to an obstetric prognosis scale: The modified SOFA scale. Ghana Med J. 2016 Sep;50(3):129-135. PMID 27752186
- [Background] Aoyama K, D'Souza R, Pinto R, Ray JG, Hill A, Scales DC, Lapinsky SE, Seaward GR, Hladunewich M, Shah PS, Fowler RA. Risk prediction models for maternal mortality: A systematic review and meta-analysis. PLoS One. 2018 Dec 4;13(12):e0208563. doi: 10.1371/journal.pone.0208563. eCollection 2018. PMID 30513118
- [Background] Oliveira-Neto AF, Parpinelli MA, Costa ML, Souza RT, Ribeiro do Valle C, Sousa MH, Cecatti JG. Prediction of Severe Maternal Outcome Among Pregnant and Puerperal Women in Obstetric ICU. Crit Care Med. 2019 Feb;47(2):e136-e143. doi: 10.1097/CCM.0000000000003549. PMID 30422862
- [Background] Vasquez DN, Estenssoro E, Canales HS, Reina R, Saenz MG, Das Neves AV, Toro MA, Loudet CI. Clinical characteristics and outcomes of obstetric patients requiring ICU admission. Chest. 2007 Mar;131(3):718-724. doi: 10.1378/chest.06-2388. PMID 17356085
- [Background] Leteurtre S, Martinot A, Duhamel A, Proulx F, Grandbastien B, Cotting J, Gottesman R, Joffe A, Pfenninger J, Hubert P, Lacroix J, Leclerc F. Validation of the paediatric logistic organ dysfunction (PELOD) score: prospective, observational, multicentre study. Lancet. 2003 Jul 19;362(9379):192-7. doi: 10.1016/S0140-6736(03)13908-6. PMID 12885479
- [Background] Vasquez DN, Das Neves AV, Vidal L, Moseinco M, Lapadula J, Zakalik G, Santa-Maria A, Gomez RA, Capalbo M, Fernandez C, Aguero-Villareal E, Vommaro S, Moretti M, Soli SB, Ballestero F, Sottile JP, Chapier V, Lovesio C, Santos J, Bertoletti F, Intile AD, Desmery PM, Estenssoro E; ProPOC Study Group. Characteristics, Outcomes, and Predictability of Critically Ill Obstetric Patients: A Multicenter Prospective Cohort Study. Crit Care Med. 2015 Sep;43(9):1887-97. doi: 10.1097/CCM.0000000000001139. PMID 26121075
- [Background] Shime N, Kageyama K, Ashida H, Tanaka Y. Application of modified sequential organ failure assessment score in children after cardiac surgery. J Cardiothorac Vasc Anesth. 2001 Aug;15(4):463-8. doi: 10.1053/jcan.2001.24983. PMID 11505351
- [Background] Estenssoro E, Kanoore Edul VS, Loudet CI, Osatnik J, Rios FG, Vazquez DN, Pozo MO, Lattanzio B, Palizas F, Klein F, Piezny D, Rubatto Birri PN, Tuhay G, Diaz A, Santamaria A, Zakalik G, Dubin A; SATISEPSIS Investigators. Predictive Validity of Sepsis-3 Definitions and Sepsis Outcomes in Critically Ill Patients: A Cohort Study in 49 ICUs in Argentina. Crit Care Med. 2018 Aug;46(8):1276-1283. doi: 10.1097/CCM.0000000000003208. PMID 29742584
- [Background] Leteurtre S, Martinot A, Duhamel A, Gauvin F, Grandbastien B, Nam TV, Proulx F, Lacroix J, Leclerc F. Development of a pediatric multiple organ dysfunction score: use of two strategies. Med Decis Making. 1999 Oct-Dec;19(4):399-410. doi: 10.1177/0272989X9901900408. PMID 10520678
- [Background] Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998 Nov;26(11):1793-800. doi: 10.1097/00003246-199811000-00016. PMID 9824069
- [Background] Shankar-Hari M, Harrison DA, Rubenfeld GD, Rowan K. Epidemiology of sepsis and septic shock in critical care units: comparison between sepsis-2 and sepsis-3 populations using a national critical care database. Br J Anaesth. 2017 Oct 1;119(4):626-636. doi: 10.1093/bja/aex234. PMID 29121281
- [Background] Ferreira FL, Bota DP, Bross A, Melot C, Vincent JL. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA. 2001 Oct 10;286(14):1754-8. doi: 10.1001/jama.286.14.1754. PMID 11594901
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239